CLINICAL TRIAL: NCT02660216
Title: A Modified Minimally Invasive Approach Towards Le Fort I Osteotomy: a Prospective Study
Acronym: MILF-I
Status: Completed | Type: Observational
Sponsor: AZ Sint-Jan AV (Other)
Responsible Party: Principal Investigator, Gwen Swennen, Maxillofacial Surgeon, MD, LDS, DMD, PhD, FEBOMFS, AZ Sint-Jan AV
Other Study IDs: BO49201525495
Record Dates: First submitted 2016-01-11; First posted 2016-01-21 (Estimated); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Jaw Abnormalities
Keywords: minimally invasive; le fort I osteotomy; 3D virtual treatment planning; accuracy
MeSH Terms: conditions — Jaw Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Nowadays, maxillary Le Fort I osteotomy is a safe and routinely performed procedure. The conventional approach is characterized by a vestibular incision extending from molar-to-molar, associated with a pterygomaxillary disjunction performed with a curved chisel. Adequate mobilization of the maxilla during Le Fort I osteotomy requires an effective separation of the maxillary tuberosity from the pterygoid plates of the sphenoid bone. However, as initially described by Precious (1991) and later by Hernandez-Alfaro (2013), a true pterygomaxillary osteotomy is not necessary to achieve successful disjunction. Furthermore, Hernandez-Alfaro combined his technique of pterygomaxillary disjunction, the so-called "Twist technique", to a minimally invasive protocol, performing the complete Le Fort I osteotomy through a 20 to 30 mm long horizontal vestibular incision. Although promising, the technique remains highly sensitive from a technical standpoint, and its true accuracy has not been comprehensively evaluated.

The purpose of this study is to present and validate a minimally invasive approach towards Le Fort I osteotomy, using a modified pterygomaxillary (PTM) disjunction technique. The primary outcome is to evaluate the accuracy of the technique using rigid voxel-based registration of the 3D virtual treatment planning and the 4 weeks postoperative CBCT images. Secondary outcomes include the surgical time necessary to complete the procedure and the presence of intraoperative and early postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients of all ages
* Patients of all genders
* A Le Fort I osteotomy is planned, as part of a bimaxillary orthognathic procedure
* The surgery is planned with 3D Virtual Treatment Planning (Maxilim v. 2.3.0.3.0.)
* The planning is transferred with 3D CAD/CAM tooth-borne splint and vertical internal bony reference landmarks
* The maxilla is repositioned first during the surgery (maxilla first sequence)

Exclusion Criteria:

* Patients not eligible according to abovementioned criteria
* Simultaneous extraction of impacted teeth 18 and/or 28
* Previous maxillary orthognathic surgery
* Previous Surgical Assisted Rapid Palatal Expansion (SARPE)
* Syndromic condition, including cleft lip and palate
* Segmental Le Fort I osteotomy
* Adjuvant Zygomatic osteotomy
* Maxillary impaction higher than 3 mm
* Maxillary advancement greater than 5 mm

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All consenting patients requiring a bimaxillary orthognathic procedure as part of their orthodontic-surgical treatment plan, and satisfying the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-11; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
accuracy of the minimally invasive approach in comparison to conventional approaches, based on 3D virtual CBCT superimposition of planning CBCT and postoperative CBCT | at 4 weeks postoperative

SECONDARY OUTCOMES:
Surgical time necessary to complete the procedure | perioperative
Intraoperative and early postoperative complications | within 4 weeks postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Gwen Swennen, Principal Investigator — Division of Maxillofacial Surgery, Department of Surgery, General Hospital Saint-John Bruges, Belgium
Locations (1):
- general hospital Saint-John Bruges, Bruges, Belgium

IPD SHARING:
Plan to Share IPD: No